CLINICAL TRIAL: NCT06852443
Title: Troubled Desire & Therapeutic Chat for Reduction of CSAM Use
Brief Title: Troubled-Desire & Therapeutic Chat for Reduction of CSAM Use (TD-CHAT)
Acronym: TD-CHAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Hannes Gieseler, Dipl.Des., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8000502101
Record Dates: First submitted 2025-02-19; First posted 2025-02-28 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Prevention; Well Being; Sexual Behavior; Behavior Change; Behavior Problems; Behavior Change Interventions; Child Sexual Abuse Material (CSAM) Consumption; Behavioral Disorder; Online Behaviour
Keywords: Child Sexual Abuse Material (CSAM) consumption; CSAM; Child Sexual Abuse; Digital online intervention; CSA; CBT; iCBT; Cognitive Behavioural Therapy; Pedophilia; chat Intervention
MeSH Terms: conditions — Sexual Behavior; Mental Disorders; Pedophilia

STUDY DESIGN:
Intervention Model Description: * Randomized
  * Multi-centre
  * Open label
  * Parallel assignment
  * Superiority
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Selfhelp+TCS (Experimental): Selfhelp modules followed by Therapist Chat Service
  Interventions: Behavioral: Selfhelp modules; Behavioral: Therapist Chat Service
- Selfhelp modules (Active Comparator): Selfhelp modules only
  Interventions: Behavioral: Selfhelp modules
- TCS only (Active Comparator): 4-6 Sessions text message-based Therapist Chat Service only
  Interventions: Behavioral: Therapist Chat Service
- Waitlist (No Intervention): Participants will remain on a waitlist for the first two weeks without receiving any kind of intervention.

INTERVENTIONS:
Behavioral: Selfhelp modules — 16 web-based structured selfhelp modules, based on CBT techniques from the Berlin Dissexuality Therapy (Beier, K. M. (2021). Pedophilia, hebephilia and sexual offending against children. The Berlin Dissexuality Therapy (BEDIT). Springer)
  Arms: Selfhelp modules; Selfhelp+TCS
Behavioral: Therapist Chat Service — Online Therapy Chat Service (TCS) based on CBT techniques from the Berlin Dissexuality Therapy (Beier, K. M. (2021). Pedophilia, hebephilia and sexual offending against children. The Berlin Dissexuality Therapy (BEDIT). Springer)
  Arms: Selfhelp+TCS; TCS only

SUMMARY:
The goal of this prospective multicentred, stratified, parallel-group superiority study is to prevent and reduce the usage of Child Sexual Abuse Material (CSAM) by a Therapist Chat Service (TCS) and Selfhelp Platform for Self-Referred Patients, mostly men with a sexual interest in children. The interventions are based on Cognitive Behavioral Therapy (CBT) principles and designed to treat the sexual behavioral disorder related with CSAM consumption.

1. Participants in the Selfhelp modules group will show a statistically significantly higher proportion of reduction in CSAM behaviours four weeks after baseline, as compared to participants in the waitlist control group.
2. Participants in the Selfhelp modules followed by TCS group will show a statistically significantly higher reduction of CSAM behaviours compared to participants in the Selfhelp-only and TCS-only groups, post-intervention.

Researchers will compare TCS-only-, Selfhelp-only-, Selfhelp + TCS- and Waiting group to see if if the interventions decrease CSAM use and improve mental well-being.

Participants will get web based selfhelp-modules and/or text-based chat intervention operated by trained therapists.

DETAILED DESCRIPTION:
The study will evaluate whether the TCS intervention and Selfhelp modules, independently or combined, effectively reduce CSAM use or risk of CSAM consumption and improve mental well-being among self-referred participants.

1. Objectives 1.1 Primary objectives

1. To compare the effectiveness in reducing CSAM behaviours between the TD only group and the waitlist group four weeks after the baseline assessment.
2. To compare the post-intervention effectiveness in reducing CSAM behaviours of the Selfhelp modules versus TCS alone and Selfhelp modules followed by TCS.

1.2 Secondary objectives

1. To assess the reduction in severity, time and self-rated risk of CSAM consumption among participants in the intervention groups (Selfhelp modules, TCS, or Selfhelp + TCS) compared to the waitlist control group, at post-intervention.
2. To compare the impact of the interventions (Selfhelp modules, TCS, or Selfhelp + TCS) on mental wellbeing, in contrast to the control group, at the end of the intervention period.
3. To evaluate the effect of the interventions (Selfhelp modules, TCS, or Selfhelp + TCS) on total sexual outlet compared with the waitlist control group after the intervention period.
4. To identify any adverse effects associated with the interventions (Selfhelp modules, TCS, or Selfhelp + TCS).

2. Hypotheses

2.1 Primary hypothesis

1. Participants in the Selfhelp-only modules group will show a statistically significantly higher proportion of reduction in CSAM behaviours four weeks after baseline, as compared to participants in the waitlist control group.
2. Participants in the Selfhelp modules followed by TCS group will show a statistically significantly higher reduction of CSAM behaviours compared to participants in the Selfhelp-only and TCS-only groups, post-intervention.

2.2 Secondary hypothesis

1. Participants in the intervention groups (Selfhelp modules, TCS, or Selfhelp + TCS) will show a statistically significant reduction in the severity, time and self-rated risk of CSAM consumption compared to participants in the waitlist control group, four weeks after the initial intervention. Among the intervention groups, it is expected that the Selfhalp + TCS group will show the greatest reduction in CSAM consumption, followed by the TCS group and then the Selfhelp-only group.
2. Participants in the intervention groups (Selfhelp modules, TCS, or Selfhelp + TCS) will show a statistically significant improvement in their mental well-being (measured using the Warwick-Edinburgh Mental Wellbeing scale). compared to participants in the waitlist control group, at post-intervention. Among the intervention groups, the Selfhelp + TCS group is expected to show the greatest improvement, followed by the TCS group, and then the Selfhelp-only group.
3. Participants in the intervention groups (Selfhelp modules, TCS, or Selfhelp + TCS) will show a statistically significant reduction in total sexual outlet (measured using a self-reported measure) compared to participants in the waitlist control group, after the intervention. Among the intervention groups, the Selfhelp + TCS group is expected to show the greatest reduction, followed by the TCS group, and then the Selfhelp-only group.
4. All intervention groups (Selfhelp modules, TCS, or Selfhelp + TCS) will experience adverse effects (psychological and emotional distress) to a similar extent, with no significant differences in the number or type of adverse effects reported. Adverse effects are expected to primarily involve mild to moderate psychological and emotional distress, such as feelings of anxiety or frustration, but are not expected to lead to severe distress or long-term harm.

3.Trial design

This is a prospective, randomised, multicentre, open-label, parallel-group, superiority trial designed to compare stratified, pair-matched CSAM users across three intervention groups and one wait-list control group, with an allocation ratio of 1:1:1:1. Following participant agreement to the terms of the study, demographic information, measures for stratified randomization, and baseline outcome data will be collected. Additionally, data collected from the four groups Selfhelp modules, TCS, Selfhelp + TCS, and waitlist) of the TD-CHAT study will be compared with data from a fifth group (waitlist + TCS) sourced from the "Scalable Technology for Online Prevention of Child Sexual Abuse and Child Sexual Abuse Materials" (STOP-CSAM) project.

ELIGIBILITY:
Inclusion Criteria:

* Adult participant (≥18 years);
* recent (last 2 weeks) CSAM use or past CSAM use and self-reported risk;
* proficiency in English, German or Spanish;
* voluntary participation and agreement to the terms of the study.

Exclusion Criteria:

* Severe neuropsychiatric comorbidities (unstable psychotic disorder, organic brain damage, diminished intellectual functioning, untreated drug or alcohol addiction);
* history of contact CSA perpetration (past or present);
* ongoing criminal investigation, trial, punishment, or probation status for online or offline CSA or CSAM use;
* current inpatient psychiatric treatment or other concurrent treatment targeting CSAM behaviours

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Child Sexual Abuse Material (RCSAM) severity | every 2 weeks for 12 weeks after onboarding
  A) Reduction in Child Sexual Abuse Material severity (RCSAM severity): A reduction in CSAM severity in the last 2 weeks, defined as the pre-post difference in highest "Combating Paedophile Information Networks in Europe" (COPINE) scale scores, with a reduction from severity levels 4 or higher to levels 3 or lower after the intervention.
Reduction in Child Sexual Abuse Material (RCSAM) time | every 2 weeks for 12 weeks after onboarding
  B) Reduction in Child Sexual Abuse Material time (RCSAM time): A 50% or greater decrease in CSAM consumption time (minutes) over the past 2 weeks. CSAM time is measured as the time (in minutes) spent consuming CSAM materials over the past 2 weeks.
Reduction in Child Sexual Abuse Material (RCSAM) risk | every 2 weeks for 12 weeks after onboarding
  C) Reduction in self-reported risk of Child Sexual Abuse Material use (RCSAM risk): A reduction in self-reported risk of CSAM use (RCSAM risk): A decrease in the risk of CSAM consumption over the last 2 weeks, defined as a pre-post decrease in self-reported risk, as measured using an adapted version of the "Sexual Child Molestation Risk Assessment" (SChiMRA+) Part A.

SECONDARY OUTCOMES:
Risk of Child Sexual Abuse Material (CSAM) consumption | baseline and 12 weeks after onboarding
  Risk of CSAM consumption: Sexual Child Molestation Risk Assessment (SchiMRA+ part A) at baseline and follow-up.
Frequency of Child Sexual Abuse Material (CSAM) consumption | baseline and every 2 weeks for 12 weeks after onboarding
  Frequency of Child Sexual Abuse Material (CSAM) consumption: Self-reported every two weeks, at baseline and follow-up.
Mental Wellbeing | baseline and every 2 weeks during 12 weeks after onboarding
  Mental wellbeing: The Warwick-Edinburgh Mental Wellbeing Scale (WEMBWS; Tennant et al., 2007). The total score is obtained by summing the score for each of the 14 items. The scoring range for each item is from 1 - 5 and the total score is from 14-70. Higher scores mean a better outcome.
  Mental wellbeing is measured over the past 2 weeks.
Total Sexual Outlet | baseline and every 2 weeks during 12 weeks after onboarding
  1. Self-reported number of orgasms achieved from masturbation using Child Sexual Abuse Material (CSAM) in the past week
  2. Self-reported number of orgasms achieved from masturbation not using CSAM in the past week
  3. Self-reported number of orgasms achieved from sexual interaction in the past week
  4. Total sexual outlet: sum of self-reported number of orgasms from masturbation (with and without using CSAM) + self-reported number of orgasms from sexual interaction.
  This outcome is measured at baseline and follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- Charité Universitätsmedizin Berlion, Berlin, Germany
- Universitat Internacional de Catalunya (UIC), Catalonia, Spain, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Landgren V, Malki K, Bottai M, Arver S, Rahm C. Effect of Gonadotropin-Releasing Hormone Antagonist on Risk of Committing Child Sexual Abuse in Men With Pedophilic Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Sep 1;77(9):897-905. doi: 10.1001/jamapsychiatry.2020.0440. PMID 32347899
- [Background] Merdian HL, Moghaddam N, Boer DP, Wilson N, Thakker J, Curtis C, Dawson D. Fantasy-Driven Versus Contact-Driven Users of Child Sexual Exploitation Material: Offender Classification and Implications for Their Risk Assessment. Sex Abuse. 2018 Apr;30(3):230-253. doi: 10.1177/1079063216641109. Epub 2016 Apr 6. PMID 27052851
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Quayle, E. (2008). The COPINE project. Irish Probation Journal, 5(9), 65-83.